CLINICAL TRIAL: NCT04982211
Title: Comparing Standard vs. Modified Reconsolidation Blockade for the Treatment of Psychological Trauma: A Randomized Controlled Trial
Brief Title: Comparing Standard vs. Modified Reconsolidation Blockade for the Treatment of Psychological Trauma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alain Brunet, Ph.D., Primary Investigator and Full Professor, Department of Psychiatry, McGill University., Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRPL-008
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Trauma and Stressor Related Disorders; Post Traumatic Stress Disorder; Acute Stress Disorder; Adjustment Disorders
Keywords: Memory Reconsolidation; Propranolol; Military personnel; Veterans; Mismatch; Efficacy
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute; Adjustment Disorders | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: This is a 2 x 2 factorial randomized controlled trial. Factor 1 is the trauma reactivation method (standard vs. mismatch trauma reactivation) and factor 2 is the study medication (propranolol vs. placebo). The design will be stratified by profession (military vs. police) and sex. After an eligibility assessment at baseline, participants meeting inclusion criteria will be randomly allocated to one of four groups with a 66.6% probability of getting enrolled in one of the two propranolol treatment groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, the investigators, therapists, outcomes assessors, and research participants will be blind to study medication allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propranolol and standard trauma memory reactivation group (Experimental): Oral propranolol will be administered 60 minutes prior to writing (Treatment 1) or reading aloud a trauma narrative.
  Interventions: Drug: Propranolol
- Placebo and standard trauma memory reactivation group (Placebo Comparator): Oral placebo will be administered 60 minutes prior to writing (Treatment 1) or reading aloud a trauma narrative.
  Interventions: Drug: Placebo
- Propranolol and mismatch trauma memory reactivation group (Active Comparator): Oral propranolol will be administered 60 minutes prior to a memory reactivation procedure involving variations in the contexts where the trauma memory reactivations occur.
  Interventions: Drug: Propranolol
- Placebo and mismatch trauma memory reactivation group (Placebo Comparator): Oral placebo will be administered 60 minutes prior to a memory reactivation procedure involving variations in the contexts where the trauma memory reactivations occur.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Oral propranolol hydrochloride capsules, dosed per participant weight
  Other Names: Teva propranolol
  Arms: Propranolol and mismatch trauma memory reactivation group; Propranolol and standard trauma memory reactivation group
Drug: Placebo — Oral placebo capsules, dosed per participant weight
  Other Names: Placebo capsules
  Arms: Placebo and mismatch trauma memory reactivation group; Placebo and standard trauma memory reactivation group

SUMMARY:
The investigators propose to examine a mismatch-based method of reconsolidation blockade for the treatment of psychological trauma in military personnel and Federal police officers. The standard reconsolidation blockade treatment (aka Reconsolidation Therapy) involves reactivating the trauma memory while under the influence of propranolol. The mismatch method of Reconsolidation Therapy will involve varying the contexts in which the weekly trauma memory retrieval will occur. This study will involve 10 visits (eligibility assessment, treatments, and follow-up visits) over a 6-month period for each participant. Treatments will be conducted once a week for a six-week period where the participant will take a dose of propranolol (or a placebo pill) 60 minutes prior to memory reactivation. The investigators hypothesize that reconsolidation blockade treatment will be as effective in treating PTSD among military personnel and Federal police officers, with the mismatch condition showing greater symptom improvement.

DETAILED DESCRIPTION:
Traumatic stress remains a treatment-refractory mental health problem characterized by symptoms of re-experiencing, avoidance, negative cognitions and affect, and hyperarousal. Due to the nature of their profession, military personnel and the Federal police officers (RCMP; Royal Canadian Mounted Police) are at a greater risk of suffering from traumatic stress. Thus, there is an important unmet need for developing novel treatments for trauma-related disorders, particularly for the military and RCMP.

Considering the pivotal role of negative emotional experiences in the development and persistence of PTSD, blocking the reconsolidation of such experiences opens the door to a novel and powerful treatment approach against this disorder. We (Brunet et al, 2018) have previously shown the efficacy of trauma memory reactivation performed under the influence of propranolol, a noradrenergic beta-receptor blocker, as a putative reconsolidation blocker, in reducing symptoms of post-traumatic stress disorder (PTSD). Although this therapeutic method was shown to be efficacious, it is hypothesized that symptomatic improvements may be increased by including a mismatch experience between what is expected during memory recall and the actual recall experience, in line with mismatch theory (Pedreira et al, 2004; see Ecker, 2015). In this study, we test the effects of a mismatch procedure by altering the context in which the trauma memory retrieval occurs. Standard and mismatch reconsolidation therapy procedures will be used to treat PTSD in military personnel and Federal police officers.

Primary objective:

• Compare the effects of Standard Reconsolidation Therapy using propranolol vs. placebo on PTSD symptoms one-week post-treatment.

Primary hypothesis:

It is predicted that propranolol administration will yield greater PTSD symptom improvement than placebo at one week following the last treatment visit.

Secondary objectives:

* Compare the effect of Standard vs. Mismatch Reconsolidation Treatment conditions on PTSD symptoms using propranolol during treatment, one-week post-treatment and at six months;
* Determine whether Reconsolidation Therapy with propranolol is associated with greater PTSD symptom reductions than placebo during treatment and at six months;
* Examine the proportion of participants rated as 'improved' based on a global clinical impression rating scale across treatment conditions;
* Examine the proportion of participants who no longer meet PTSD diagnostic criteria at one-week post-treatment and follow-up according to treatment condition;
* Explore the effect of the treatment on depressive symptoms, dissociative symptoms, complex PTSD symptomatology, and quality of life;
* Examine the effect of treatment condition on drop-outs and relapse rates;

Procedures

To accomplish the study objectives, the investigators will employ a randomized, double-blind, placebo-controlled trial and use standardized, repeated dependent measures of change at each treatment visit, as well as at one-week, 3-month and 6-month post-treatment visits). At each treatment session, participants will be asked recall their traumatic memory with the help of a trauma narrative under the influence of propranolol or a placebo. Recall will occur using a standard reconsolidation or mismatch protocol. Four treatment conditions will be defined, as follows:

* Group 1: Standard trauma memory reactivation + propranolol;
* Group 2: Standard trauma reactivation + placebo;
* Group 3: Modified trauma reactivation + propranolol;
* Group 4: Modified trauma reactivation + placebo.

As a means to favor recruitment, the current study will use an unbalanced sampling design. We will randomize 50 participants per cell in each of two active treatment groups and 25 participants per cell in the two placebo groups. Approximately 4 sites will be involved in recruiting participants for the study: one in the US, with the remaining sites in Canada. We are targeting 150 study participants with the aim of obtaining 121 treatment completers, taking into account an approximate 20% attrition rate.

The protocol will involve 10 study visits over a 6-month period. The first two visits will serve to obtain consent, establish the PTSD diagnosis, and determine eligibility. Treatments will occur once a week for 6 weeks. The standard reconsolidation therapy procedure will involve having participants write or read a summary of their traumatic experience under the influence of propranolol. The mismatch reconsolidation therapy condition will involve changing the way the trauma narrative is used to reactivate the trauma memory at each visit . Participants will not be informed in advance of the mismatch procedures. Follow-up assessments for all participants will be conducted one week post-treatment, as well as at three- and six-months after study entry.

Statistical Analyses. It is hypothesized that both standard and mismatch therapy conditions under propranolol will show greater improvements than with placebo. However, it is the mismatch therapy condition using propranolol is expected to yield significantly greater improvements in PTSD symptoms relative to the other three conditions. All data will be tested using mixed effects statistical models.

ELIGIBILITY:
Inclusion Criteria:

(i) Male or female 18-65 years old;

(ii) Individuals who are either:

* Employed full-time as part of the Canadian or US military forces or the RCMP;
* On leave of absence from Canadian or US military forces, or the RCMP;
* Veterans of the Canadian or US military forces or the RCMP;

(iii) Evidence of a personally signed and dated informed consent form;

(iv) Individuals suffering from occupationally related PTSD, as defined by the DSM-5, for 6 consecutive months or more.

(v) Females of childbearing potential willing to use contraception for the duration of the treatment period of the study.

Exclusion Criteria:

(i) Basal systolic blood pressure < 100 mm Hg;

(ii) Basal heart rate < 50 BPM;

(iii) Medical conditions contraindicating the administration of propranolol or beta blockers

(iv) A known hypersensitivity to propranolol or any of the study product or placebo ingredients;

(v) Clinically significant lactose intolerance;

(vi) Use of medication that involves unwanted interactions with propranolol including but not limited to other beta-blockers, anti-arrhythmic medications, and calcium channel blockers;

(vii) Current use of propranolol;

(viii) Pregnant or breast-feeding women;

(ix) Individuals with borderline personality, bipolar disorder, psychosis;

(x) Current DSM-5 substance dependence;

(xi) Active suicidal ideations, as demonstrated by a response of 2 or 3 on item 7 of the Beck Depression Inventory - Short Form;

(xii) A score below 'moderately ill' on the severity scale of the Clinical Global Impression scale;

(xiii) Participating in active litigation related to the traumatic event (Veterans Affairs Canada claims are permitted, excluding judicial claims);

(xiv) Strong dissociative tendencies, as evidenced by the Dissociative Experience Scale (8-item version, DES-T);

(xv) Suspected or confirmed traumatic brain injury during the last 24 months;

(xvi) Understanding neither English nor French;

(xvii) Participants who receive exposure-based cognitive-behavioral therapy during the treatment phase of the study;

(xviii) Presence of any medical condition that in the opinion of the investigator may compromise patient safety or study objectives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic Checklist for the Diagnostic and Statistical Manual for Mental Disorders - 5th edition (PCL-5) scores | Questionnaire administered at weeks 0 and 7
  Change from baseline (week 0) to week 7 in PCL-5 scores

SECONDARY OUTCOMES:
Post-traumatic Checklist for the Diagnostic and Statistical Manual for Mental Disorders - 5th edition (PCL-5) scores | Questionnaire administered at weeks 0, 1, 2, 3, 4, 5, 6, 13 and 26
  Changes from baseline in PCL-5 scores during treatment and at weeks 13 and 26
Beck Depression Inventory (BDI) scores | Questionnaire administered at weeks 0, 1, 2, 3, 4 , 5, 6, 7, 13 and 26
  Changes from baseline in BDI scores during treatment and at week 26
Clinical Global Impression-Improvement (CGI-I) scores | Questionnaire administered at weeks 0, 7 and 26
  Absolute CGI-I scores
Mini Psychiatric Interview, version 7 (MINI-7) | Questionnaire administered at weeks 0, 7 and 26
  Proportion of participants who no longer meet PTSD diagnostic criteria at Weeks 7 and 26.
Social Functioning Questionnaire (QFS) | Questionnaire administered at weeks 0, 7, and 26
  Changes from baseline in QFS scores
World Health Organization - Quality of Life BREF | Questionnaire administered at weeks 0, 7, and 26
  Changes from baseline in World Health Organization - Quality of Life BREF scores
Dissociative Experiences Scale (DES-T) | Questionnaire administered at week 0.
  Changes from baseline in DES-T scores
International Trauma Questionnaire (ITQ) | Questionnaire administered at baseline and weeks 0, 7, and 26
  Changes from baseline in ITQ scores

CONTACTS AND LOCATIONS:
Overall Officials: Alain Brunet, Ph.D., Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunet A, Saumier D, Liu A, Streiner DL, Tremblay J, Pitman RK. Reduction of PTSD Symptoms With Pre-Reactivation Propranolol Therapy: A Randomized Controlled Trial. Am J Psychiatry. 2018 May 1;175(5):427-433. doi: 10.1176/appi.ajp.2017.17050481. Epub 2018 Jan 12. PMID 29325446
- [Background] Ecker B. Memory reconsolidation understood and misunderstood. International Journal of Neuropsychotherapy. 2015; 3(1): 2-46.
- [Background] Cheymol G. Clinical pharmacokinetics of drugs in obesity. An update. Clin Pharmacokinet. 1993 Aug;25(2):103-14. doi: 10.2165/00003088-199325020-00003. PMID 8403734
- [Background] Sevenster D, Beckers T, Kindt M. Prediction error governs pharmacologically induced amnesia for learned fear. Science. 2013 Feb 15;339(6121):830-3. doi: 10.1126/science.1231357. PMID 23413355
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Fliess JL. The Design and Analysis of Clinical Experiments. New York: John Wiley,1986.
- [Background] Desmeules J. Interations médicamenteuses et cytochromes P450. Pharma-Flash, 2002. 29(4): 13-16.
- [Background] Mackinnon A. The use and reporting of multiple imputation in medical research - a review. J Intern Med. 2010 Dec;268(6):586-93. doi: 10.1111/j.1365-2796.2010.02274.x. Epub 2010 Sep 10. PMID 20831627
- [Background] Benjamini, Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. Journal of the Royal Statistical Society.1995; Series B (Methodological): 289-300.
- [Background] Pedreira ME, Perez-Cuesta LM, Maldonado H. Mismatch between what is expected and what actually occurs triggers memory reconsolidation or extinction. Learn Mem. 2004 Sep-Oct;11(5):579-85. doi: 10.1101/lm.76904. PMID 15466312